CLINICAL TRIAL: NCT01982331
Title: Reactogenicity, Safety and Immunogenicity of a Live Monovalent A/17/California/66/395 (H2N2)Influenza Vaccine
Brief Title: Reactogenicity, Safety and Immunogenicity of a Live Monovalent A/17/CALIFORNIA/66/395 (H2N2) Influenza Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PATH (Other)
Collaborators: Ministry of Health, Russian Federation (Other Government); Institute of Experimental Medicine, Russia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LAIV-H2N2-01
Record Dates: First submitted 2013-10-30; First posted 2013-11-13 (Estimated); Results first posted 2019-02-06 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Influenza
Keywords: H2N2; vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LAIV H2N2 vaccine (Experimental): LAIV H2N2 vaccine A/17/California/66/395 (H2N2) live monovalent influenza vaccine delivered intranasally 2 doses 1 month apart
  Interventions: Biological: LAIV H2N2
- Placebo (Placebo Comparator): Placebo is composed of a lyophilizate containing the same concentrations of stabilizers as LAIV vaccine. It is prepared onsite in an identical fashion to the vaccine and delivered intranasally.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: LAIV H2N2 — vaccine is delivered intranasally, .25 cc to each nostril at day 0 and day 28
  Other Names: Monovalent A/17/California/66/395 (LAIV H2N2) vaccine
  Arms: LAIV H2N2 vaccine
Other: Placebo — placebo delivered intranasally. .25cc to each nostril at day 0 and day 28
  Arms: Placebo

SUMMARY:
This is a phase I study to evaluate the safety of a vaccine to protect against influenza viruses of the H2N2 subtype. A total of 40 adults will be enrolled and receive two doses of vaccine or placebo one month apart.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the safety profile of two intranasal doses of LAIV A/17/California/66/395 (H2N2) in healthy adults in Russia. A(H2N2) viruses which are antigenically similar to the pandemic strain A/Singapore/1/57, continue to circulate in domestic and wild bird populations, as confirmed by routine moni¬toring of avian influenza viruses.

40 adults aged 18-40 will be enrolled. They will be randomized to receive vaccine or placebo. Blood and urine will be collected during the week following each vaccination and before the next vaccination to monitor safety. Blood samples will also be collected at several timepoints to assess the volunteer's immune response to the vaccine. The total duration of the study is 16 weeks for each volunteer.

ELIGIBILITY:
Inclusion Criteria:

* Legal male or female adult aged 18 through 40 years
* Literate and willing to provide written informed consent.
* A signed informed consent.
* Free of obvious health problems, as established by medical history and screening evaluations, including physical examination.
* Capable and willing to complete diary cards and willing to return for all follow-up visits
* Willing to comply with the rules of isolation unit (including willing and able to take oseltamivir influenza antiviral medication, should that be recommended by study physician).
* For females, willing to take reliable birth control measures through day 56.

Exclusion Criteria:

* Participation in another clinical trial involving any therapy within the previous three months or planned enrollment in such a trial during trial period.
* Receipt of any non-study vaccine within four weeks prior to enrollment or refusal to postpone receipt of such vaccines until four weeks after study completion.
* Practice of nasal irrigation on a regular basis within the past six months or has engaged in nasal irrigation within two weeks prior to enrollment.
* Recent history of frequent nose bleeds (>5 within the past year).
* Clinically relevant abnormal paranasal anatomy.
* Recent history (within the past month) of rhino or sinus surgery, or surgery for any traumatic injury of the nose.
* Current or recent (within two weeks of enrollment) acute respiratory illness with or without fever.
* Other acute illness at the time of study enrollment.
* Receipt of immune globulin or other blood products within three months prior to study enrollment or planned receipt during period of subject participation in the study.
* Chronic administration (defined as more than 14 consecutively-prescribed days) of immunosuppressants and/or other immune-modulating therapy within six months prior to study enrollment.
* Participation in any previous trial of any H2N2 containing influenza vaccine.
* History of asthma.
* Hypersensitivity after previous administration of any influenza vaccine.
* History of wheezing after past receipt of any live influenza vaccine.
* Other adverse event (AE) following immunization (body temperature more than 40°C, collapse, non-febrile seizures, anaphylaxis), at least possibly related to previous receipt of any vaccine (not only influenza).
* Suspected or known hypersensitivity to any study vaccine components, including chicken or egg protein.
* Seasonal (autumnal) hypersensitivity to the natural environment
* Acute or chronic clinically significant pulmonary, cardiovascular, hepatic, metabolic, neurologic, psychiatric or renal functional abnormality, as determined by medical history, physical examination or clinical laboratory screening tests, which in the opinion of the investigator, might interfere with the study objectives. Subjects with physical examination findings or clinical laboratory screening results which would be graded 2 or higher on the AE severity grading scale (see Attachments) will be excluded from entry into the study and will be excluded from receipt of dose two of study vaccine or placebo.
* History of leukemia or any other blood or solid organ cancer.
* History of thrombocytopenic purpura or known bleeding disorder.
* History of seizures.
* Known or suspected immunosuppressive or immunodeficient condition of any kind, including HIV infection.
* Known chronic hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
* Known tuberculosis infection or evidence of previous tuberculosis exposure.
* History of chronic alcohol abuse and/or illegal drug use.
* Claustrophobia or sociophobia.
* Pregnancy or lactation.
* Any condition that, in the opinion of the investigator, would increase the health risk to the subject if participates in the study or would interfere with the evaluation of the study objectives.
* Allergic, including anaphylactic, reactions to the introduction of any vaccines (not only influenza) in the subject's medical history

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2013-10; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oleg I Kiselev, Ph.D., Principal Investigator — Research Institute of Influenza; Jorge E Flores, MD, Ph.D., Study Director — PATH
Locations (1):
- Research Institute of Influenza, Saint Petersburg, Russia

REFERENCES:
- [Derived] Rak A, Donina S, Zabrodskaya Y, Rudenko L, Isakova-Sivak I. Cross-Reactivity of SARS-CoV-2 Nucleocapsid-Binding Antibodies and Its Implication for COVID-19 Serology Tests. Viruses. 2022 Sep 14;14(9):2041. doi: 10.3390/v14092041. PMID 36146847
- [Derived] Kiseleva I, Dubrovina I, Fedorova E, Larionova N, Isakova-Sivak I, Bazhenova E, Pisareva M, Kuznetsova V, Flores J, Rudenko L. Genetic stability of live attenuated vaccines against potentially pandemic influenza viruses. Vaccine. 2015 Dec 8;33(49):7008-14. doi: 10.1016/j.vaccine.2015.09.050. Epub 2015 Oct 2. PMID 26432909

RESULTS

PARTICIPANT FLOW:
Period: Received Vaccination 1
Arm/Group | LAIV H2N2 Vaccine | Placebo
Started | 28 | 10
Completed | 28 | 10
Not Completed | 0 | 0
Period: Received Vaccination 2
Arm/Group | LAIV H2N2 Vaccine | Placebo
Started | 28 | 10
Completed | 27 | 7
Not Completed | 1 | 3
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1
Period: Completed Study (Day 112)
Arm/Group | LAIV H2N2 Vaccine | Placebo
Started | 27 | 7
Completed | 25 | 7
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LAIV H2N2 Vaccine | Placebo | Total
Number analyzed (Participants) | 28 | 10 | 38
Age, Continuous [Mean (Full Range); unit: years] | 28.0 [18 to 40] | 26.2 [18 to 40] | 27.6 [18 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 3 | 15
  Male | 16 | 7 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 28 | 10 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 28 | 10 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Russia | 28 | 10 | 38

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Immediate Reactions
Description: Measured as observed by study staff or reported by the subject to study staff whether related or not related.
Time Frame: 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | LAIV H2N2 Vaccine | Placebo
Number analyzed (Participants) | 28 | 10
Participants
  Vaccination 1: Yes | 0 | 0
  Vaccination 1: No | 28 | 10
  Vaccination 2: Yes | 0 | 0
  Vaccination 2: No | 28 | 10

2. Primary Outcome: Percentage of Subjects With Solicited Local and Systemic Reactions After Vaccination 1
Description: Adverse events commonly associated with intranasal vaccination occurring greater than two hours after administration of any dose of study vaccine or placebo through 6 days following any dose, measured as observed by study staff or reported by the subject to study staff. Solicited local reactions included: dryness of the nose, nose bleeds, ticklish nose, nasal congestion, runny nose, ticklish throat, catarrhal nasopharynx. Solicited systemic reactions included: body temperature, feverishness/subjective fever, chills, cough, difficulty breathing, sore throat, headache, confusion, convulsions/seizures, fatigue/malaise, joint aches, muscle aches, pink or red eyes, draining eyes, swollen eyelids, ear pain or discharge, rash, abdominal pain, diarrhea, vomiting.
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | LAIV H2N2 Vaccine | Placebo
Number analyzed (Participants) | 28 | 10
Participants
  Any solicited local or systemic reaction: Yes | 13 | 5
  Any solicited local or systemic reaction: No | 15 | 5
  Any solicited local reaction: Yes | 4 | 2
  Any solicited local reaction: No | 24 | 8
  Any solicited systemic reaction: Yes | 13 | 4
  Any solicited systemic reaction: No | 15 | 6

3. Primary Outcome: Percentage of Subjects With Solicited Local and Systemic Reactions After Vaccination 2
Description: as for outcome 2
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | LAIV H2N2 Vaccine | Placebo
Number analyzed (Participants) | 28 | 10
Participants
  Any solicited local or systemic reaction: Yes | 9 | 2
  Any solicited local or systemic reaction: No | 19 | 8
  Any solicited local reaction: Yes | 0 | 0
  Any solicited local reaction: No | 28 | 10
  Any solicited systemic reaction: Yes | 9 | 2
  Any solicited systemic reaction: No | 19 | 8

4. Primary Outcome: Percentage of Subjects With Unsolicited Adverse Events After Vaccination 1
Description: All other adverse events (including unsolicited events and abnormal laboratory parameters) occurring during the 6 days following any dose, measured as observed by study staff or reported by the subject to study staff.
Time Frame: 7 days following each vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | LAIV H2N2 Vaccine | Placebo
Number analyzed (Participants) | 28 | 10
Participants
  Unrelated to vaccination: Yes | 15 | 7
  Unrelated to vaccination: No | 13 | 3
  Related to vaccination: Yes | 16 | 5
  Related to vaccination: No | 12 | 5

5. Primary Outcome: Percentage of Subjects With Unsolicited Adverse Events After Vaccination 2
Description: as for outcome 4
Time Frame: 7 days following each vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | LAIV H2N2 Vaccine | Placebo
Number analyzed (Participants) | 28 | 10
Participants
  Unrelated to vaccination: Yes | 19 | 6
  Unrelated to vaccination: No | 9 | 4
  Related to vaccination: Yes | 19 | 4
  Related to vaccination: No | 9 | 6

6. Secondary Outcome: Percentage of Subjects With Seroconversion for Serum Hemagglutination Inhibition (HAI) Antibodies
Description: Defined as a 4-fold or higher response from baseline (day 0), 28 days after each vaccination and after 112 days.
Time Frame: Day 28, Day 56 and Day 112
Population: Subjects that received each vaccination (vaccination 1 for day 28, vaccination 2 for days 56 and 112), did not withdraw from the study, and that had viable immunologic data.
Measure: Count of Participants; unit: Participants
Arm/Group | LAIV H2N2 Vaccine | Placebo
Number analyzed (Participants) | 25 | 7
Participants
  Day 28: Yes | 4 | 0
  Day 28: No | 21 | 7
  Day 56: Yes | 8 | 0
  Day 56: No | 17 | 7
  Day 112: Yes | 15 | 0
  Day 112: No | 10 | 7

7. Secondary Outcome: Percentage of Subjects With Seroconversion for Serum Neutralizing Antibodies
Description: Defined as a 4-fold or higher response from baseline (day 0), 28 days after each vaccination and after 112 days. Measured by microneutralization assay.
Time Frame: Day 28, Day 56 and Day 112
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | LAIV H2N2 Vaccine | Placebo
Number analyzed (Participants) | 25 | 7
Participants
  Day 28: Yes | 8 | 1
  Day 28: No | 17 | 6
  Day 56: Yes | 10 | 1
  Day 56: No | 15 | 6
  Day 112: Yes | 11 | 1
  Day 112: No | 14 | 6

8. Secondary Outcome: Percentage of Subjects With Seroconversion for Serum Immunoglobulin A Antibodies
Description: Defined as a 4-fold or higher response from baseline (day 0), 28 days after each vaccination and after 112 days. Measured by enzyme-linked immunosorbent assay (ELISA).
Time Frame: Day 28, Day 56 and Day 112
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | LAIV H2N2 Vaccine | Placebo
Number analyzed (Participants) | 25 | 7
Participants
  Day 28: Yes | 2 | 0
  Day 28: No | 23 | 7
  Day 56: Yes | 13 | 0
  Day 56: No | 12 | 7
  Day 112: Yes | 12 | 0
  Day 112: No | 13 | 7

9. Secondary Outcome: Percentage of Subjects With Seroconversion for Serum Immunoglobulin G Antibodies
Description: as for outcome 8
Time Frame: Day 28, Day 56 and Day 112
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | LAIV H2N2 Vaccine | Placebo
Number analyzed (Participants) | 25 | 7
Participants
  Day 28: Yes | 0 | 0
  Day 28: No | 25 | 7
  Day 56: Yes | 1 | 0
  Day 56: No | 24 | 7
  Day 112: Yes | 2 | 0
  Day 112: No | 23 | 7

10. Secondary Outcome: Percentage of Subjects With Seroconversion for Secretory Immunoglobulin A Antibodies From Nasal Mucosa
Description: Defined as a 4-fold or higher response from baseline (day 0), 28 days after each vaccination.
Time Frame: Day 28 and Day 56
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | LAIV H2N2 Vaccine | Placebo
Number analyzed (Participants) | 25 | 7
Participants
  Day 28: Yes | 6 | 0
  Day 28: No | 19 | 7
  Day 56: Yes | 10 | 0
  Day 56: No | 15 | 7

11. Secondary Outcome: Percentage of Subjects With Seroconversion for Secretory Immunoglobulin A Antibodies Detected in Saliva Specimens
Description: Defined as a 4-fold or higher response from baseline (day 0), 28 days after each vaccination.
Time Frame: Day 28 and Day 56
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | LAIV H2N2 Vaccine | Placebo
Number analyzed (Participants) | 25 | 7
Participants
  Day 28: Yes | 3 | 0
  Day 28: No | 22 | 7
  Day 56: Yes | 9 | 0
  Day 56: No | 16 | 7

12. Secondary Outcome: Percentage of Subjects Shedding Influenza A Virus Using Nasal Swab
Description: Detected by real-time reverse transcriptase polymerase chain reaction. Specimens were collected prior to each vaccination and 7 days post-vaccination.
Time Frame: Days 0-6 and Days 28-34
Measure: Count of Participants; unit: Participants
Arm/Group | LAIV H2N2 Vaccine | Placebo
Number analyzed (Participants) | 27 | 7
Participants
  Day 0 pre-dose: Negative | 27 | 7
  Day 0 pre-dose: Positive | 0 | 0
  Day 1: Negative | 6 | 7
  Day 1: Positive | 21 | 0
  Day 2: Negative | 17 | 7
  Day 2: Positive | 10 | 0
  Day 3: Negative | 23 | 7
  Day 3: Positive | 4 | 0
  Day 4: Negative | 25 | 7
  Day 4: Positive | 2 | 0
  Day 5: Negative | 27 | 7
  Day 5: Positive | 0 | 0
  Day 6: Negative | 27 | 7
  Day 6: Positive | 0 | 0
  Day 28 pre-dose: Negative | 27 | 7
  Day 28 pre-dose: Positive | 0 | 0
  Day 29: Negative | 7 | 7
  Day 29: Positive | 20 | 0
  Day 30: Negative | 25 | 7
  Day 30: Positive | 2 | 0
  Day 31: Negative | 27 | 7
  Day 31: Positive | 0 | 0
  Day 32: Negative | 27 | 7
  Day 32: Positive | 0 | 0
  Day 33: Negative | 27 | 7
  Day 33: Positive | 0 | 0
  Day 34: Negative | 27 | 7
  Day 34: Positive | 0 | 0

13. Secondary Outcome: Percentage of Subjects Shedding Influenza Virus Subtype Using Nasal Swab
Description: as for outcome 12
Time Frame: Days 0-6 and Days 28-34
Measure: Count of Participants; unit: Participants
Arm/Group | LAIV H2N2 Vaccine | Placebo
Number analyzed (Participants) | 27 | 7
Participants
  Day 0 pre-dose: Negative | 27 | 7
  Day 0 pre-dose: H2 | 0 | 0
  Day 1: Negative | 7 | 7
  Day 1: H2 | 20 | 0
  Day 2: Negative | 18 | 7
  Day 2: H2 | 9 | 0
  Day 3: Negative | 23 | 7
  Day 3: H2 | 4 | 0
  Day 4: Negative | 26 | 7
  Day 4: H2 | 1 | 0
  Day 5: Negative | 27 | 7
  Day 5: H2 | 0 | 0
  Day 6: Negative | 27 | 7
  Day 6: H2 | 0 | 0
  Day 28 pre-dose: Negative | 27 | 7
  Day 28 pre-dose: H2 | 0 | 0
  Day 29: Negative | 7 | 7
  Day 29: H2 | 20 | 0
  Day 30: Negative | 25 | 7
  Day 30: H2 | 2 | 0
  Day 31: Negative | 27 | 7
  Day 31: H2 | 0 | 0
  Day 32: Negative | 27 | 7
  Day 32: H2 | 0 | 0
  Day 33: Negative | 27 | 7
  Day 33: H2 | 0 | 0
  Day 34: Negative | 27 | 7
  Day 34: H2 | 0 | 0

14. Secondary Outcome: Percentage of Subjects Shedding Influenza A Virus Using Throat Swab
Description: as for outcome 12
Time Frame: Days 0-6 and Days 28-34
Measure: Count of Participants; unit: Participants
Arm/Group | LAIV H2N2 Vaccine | Placebo
Number analyzed (Participants) | 27 | 7
Participants
  Day 0 pre-dose: Negative | 27 | 7
  Day 0 pre-dose: Positive | 0 | 0
  Day 1: Negative | 27 | 7
  Day 1: Positive | 0 | 0
  Day 2: Negative | 25 | 7
  Day 2: Positive | 2 | 0
  Day 3: Negative | 27 | 7
  Day 3: Positive | 0 | 0
  Day 4: Negative | 27 | 7
  Day 4: Positive | 0 | 0
  Day 5: Negative | 27 | 7
  Day 5: Positive | 0 | 0
  Day 6: Negative | 27 | 7
  Day 6: Positive | 0 | 0
  Day 28 pre-dose: Negative | 27 | 7
  Day 28 pre-dose: Positive | 0 | 0
  Day 29: Negative | 25 | 7
  Day 29: Positive | 2 | 0
  Day 30: Negative | 26 | 7
  Day 30: Positive | 1 | 0
  Day 31: Negative | 27 | 7
  Day 31: Positive | 0 | 0
  Day 32: Negative | 27 | 7
  Day 32: Positive | 0 | 0
  Day 33: Negative | 27 | 7
  Day 33: Positive | 0 | 0
  Day 34: Negative | 27 | 7
  Day 34: Positive | 0 | 0

15. Secondary Outcome: Percentage of Subjects Shedding Influenza Virus Subtype Using Throat Swab
Description: as for outcome 12
Time Frame: Days 1-6 and Days 29-34
Measure: Count of Participants; unit: Participants
Arm/Group | LAIV H2N2 Vaccine | Placebo
Number analyzed (Participants) | 27 | 7
Participants
  Day 1: Negative | 27 | 7
  Day 1: H2 | 0 | 0
  Day 2: Negative | 27 | 7
  Day 2: H2 | 0 | 0
  Day 3: Negative | 27 | 7
  Day 3: H2 | 0 | 0
  Day 4: Negative | 27 | 7
  Day 4: H2 | 0 | 0
  Day 5: Negative | 27 | 7
  Day 5: H2 | 0 | 0
  Day 6: Negative | 27 | 7
  Day 6: H2 | 0 | 0
  Day 29: Negative | 25 | 7
  Day 29: H2 | 2 | 0
  Day 30: Negative | 26 | 7
  Day 30: H2 | 1 | 0
  Day 31: Negative | 27 | 7
  Day 31: H2 | 0 | 0
  Day 32: Negative | 27 | 7
  Day 32: H2 | 0 | 0
  Day 33: Negative | 27 | 7
  Day 33: H2 | 0 | 0
  Day 34: Negative | 27 | 7
  Day 34: H2 | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 days following either dose for non-serious adverse events, and 4 weeks after either dose for serious adverse events.
Arm/Group | LAIV H2N2 Vaccine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/10
Other Adverse Events (participants affected / at risk) | 26/28 | 9/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LAIV H2N2 Vaccine (N=28) | Placebo (N=10)
Ear congestion (Ear and labyrinth disorders) | 1 | 0
Fatigue (General disorders) | 1 | 1
Pyrexia (General disorders) | 2 | 2
Bronchitis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 2
Periodontitis (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 3 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 0
Blood bicarbonate increased (Investigations) | 2 | 3
Blood bilirubin increased (Investigations) | 6 | 2
Blood calcium increased (Investigations) | 4 | 1
Blood creatinine increased (Investigations) | 2 | 1
Blood glucose increased (Investigations) | 7 | 2
Blood urea increased (Investigations) | 2 | 0
Eosinophil count increased (Investigations) | 4 | 0
Haemoglobin increased (Investigations) | 3 | 0
Lymphocyte count decreased (Investigations) | 5 | 2
Lymphocyte count increased (Investigations) | 21 | 6
Mean cell haemoglobin concentration increased (Investigations) | 3 | 2
Monocyte count increased (Investigations) | 10 | 2
Neutrophil count decreased (Investigations) | 13 | 6
Neutrophil count increased (Investigations) | 1 | 1
Protein total decreased (Investigations) | 3 | 2
Red blood cell count decreased (Investigations) | 0 | 1
Red blood cell count increased (Investigations) | 1 | 0
Red blood cell sedimentation rate increased (Investigations) | 4 | 2
White blood cell count increased (Investigations) | 0 | 1
Headache (Investigations) | 1 | 1
Nasal congestion (Investigations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No